CLINICAL TRIAL: NCT06835673
Title: PREVALENCE OF ANXIETY AND DEPRESSION AMONG FAMILY MEMBERS OF ICU PATIENTS IN A TERTIARY-LEVEL HOSPITAL IN NEPAL: A PROSPECTIVE OBSERVATIONAL STUDY
Brief Title: The ICU is a Complex Setting Where Critically Ill Patients Are Treated, Impacting Caregivers' Mental Health, Leading to Anxiety and Depression .we Aim to Identify the Prevalence of Anxiety and Depression Among Family Members of ICU Patients in a Tertiary-Level Hospital in Nepal
Acronym: HADS
Status: Completed | Type: Observational
Sponsor: Tribhuvan University Teaching Hospital, Institute Of Medicine. (Other)
Responsible Party: Principal Investigator, Sadikshya Regmi, Doctor, Tribhuvan University Teaching Hospital, Institute Of Medicine.
Other Study IDs: 202(6-11)E2; PROFF DR BISHWAS PRADHAN (Other: TUTH)
Record Dates: First submitted 2025-02-14; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Anxiety Disorder/Anxiety State
Keywords: anxiety and depression; FAMILY MEMBERS; CRITICALLY ILL; ICU; HADS
MeSH Terms: conditions — Anxiety Disorders; Depression; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- interview of caretaker/ visitors of the patients who are admitted to the ICU for more than 48 hours: a validated tool of anxiety and depression HADS ( HOSPITAL ANXIETY AND DEPRESSION SCORE) used in a structured way to interview the caretaker/visitors of the critically ill patients admitted in ICU

SUMMARY:
a prospective observational study conducted in ICU of tertiary hospital under the guidance of mentors of department of critical care medicine TUTH to identify the Prevalence of Anxiety and Depression Among Family Members of ICU Patients in a Tertiary-Level Hospital in Nepal

DETAILED DESCRIPTION:
Rationale:

The Intensive Care Unit (ICU) is a demanding environment designed to care for critically ill patients requiring constant medical attention and specialized resources. Admission to the ICU is extremely stressful for both patients and their families, leading to considerable physical and mental stress which can manifests as anxiety and depression. Understanding the prevalence of these conditions and their association with unmet needs is crucial for developing targeted interventions.

Study objective:

Design: A prospective cross sectional descriptive study design Duration: August-Nov 2024 Place: Intensive care units (ICUs) of the Department of Critical Care Medicine, Tribhuvan University Teaching Hospital (TUTH) and Intensive care units (ICUs) of MMC

Introduction The Intensive Care Unit (ICU) is a critical care environment designed to provide continuous and intensive medical attention to patients with severe and life-threatening conditions. The complex medical interventions and the high-stress environment within the ICU have significant psychological impacts not only on the patients but also on their family members. The emotional burden experienced by relatives during a loved one's ICU stay is profound and often manifests as anxiety and depression.

Relatives of ICU patients frequently report high levels of stress, anxiety, and depression due to the uncertain prognosis and the intimidating ICU environment. Despite the recognition of these emotional challenges, there is a lack of comprehensive studies that quantify the prevalence of anxiety and depression among family members and correlate these conditions with their unmet needs during the ICU stay. Addressing these gaps is essential for developing effective support strategies.

Study variables Baseline characteristics Age Gender Diagnosis Marital status APACHE II score Calculated mortality rate Illness (acute or chronic) Planned / unplanned admission Admission from ED/ ward Interventions done to the patients Intubation and mechanical ventilation Hemodialysis catheter / CRRT Chest tube insertion Foley's catheterization Nasogastric tube insertion Central line insertion Surgical drain Restraints Tracheostomy

Visitor Baseline Characteristics:

Gender Age Education Marital status Relationship with the patient Previous ICU hospitalizations in the family Residence with the patient Number of visits per day Occupation status

Expected time and duration of the study Sample size of 110 will be collected.

Tools and techniques for data collection The tools that will be used in this study include The Hospital Anxiety and Depression Scale (HADS), modified in the Nepali version All data will be recorded using pre-formed proformas.

Management protocol of patients/participants Family members of all adult patients who are equal to or >18 years of age will be included in the study.

Patients should be admitted in the ICU for at least 48 hours. Visitors who are next to the kin ( nearest ) care taker will be chosen for the interview.

As a routine care of the ICU ,family members have fixed visiting hours in the ICU.

The one to be interviewed will have to visit the ICU and his admitted family member at least once in these 48 hours.

Also, as routine care Family members of the admitted patients are counselled by the doctors on duty at least once a day regarding the ware bouts of the patients and further if required.

Family members are also counselled by the assigned bed side nurse of the patient about the visiting hours and orientation regarding ICU rules and requirements.

Family members who have visited his patient once and who has been once counselled by the assigned nurse and the duty doctor at least once will be interviewed by the interviewer.

Interview can be taken at any time of the day as per the convenience or the member for interview or the interviewer.

Patients' demographics and baseline characteristics will be taken from the ICU data.

The tubes and catheters that the patients had during the family member's visit were recorded to detect how these interventions affected the family member's mood state APACHE 2 score will be calculated of the 1st 24 hours of admission. An informed written consent will be obtained from the interviewee before the commencement of the interview.

Family member's characteristics will be obtained by the interview. HADS questionnaire will be used as the tool for assessing the anxiety and depression amongst family members.

Family member will be given the option of either self-assessing the questionnaire or if not able to read and write will be directed by the interviewer himself/ herself by reading out the questionnaire.

HADS questionnaires is attached at the end of the proforma. No cameras , voice tape or video will be recorded. Baseline characteristics Age Gender Diagnosis Marital status APACHE II score Calculated mortality rate Illness (acute or chronic) Planned / unplanned admission Admission from ED/ ward Interventions done to the patients Intubation and mechanical ventilation Hemodialysis catheter / CRRT Chest tube insertion Foley's catheterization Nasogastric tube insertion Central line insertion Surgical drain Restraints Tracheostomy

Visitor Baseline Characteristics:

Gender Age Education Marital status Relationship with the patient Previous ICU hospitalizations in the family Day of hospitalization Residence with the patient Number of visits per day Occupation status

ELIGIBILITY:
Inclusion Criteria:

Family members aged 18 and above Family members of patients who have been admitted to the ICU for more than 48 hours.

-

Exclusion Criteria:

Family members who refuse to give consent. Unable to understand Nepali language.

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Family members aged 18 and above Family members of patients who have been admitted to the ICU for more than 48 hours.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Prevalence of Anxiety and Depression Among Family Members of ICU Patients in a Tertiary-Level Hospital in Nepal | 4 months
  caretaker visitors of the critically ill patients admitted in ICU of TUTH were interviewed using a validated score HADS to see the prevalence of anxiety and depression amongst them.

CONTACTS AND LOCATIONS:
Locations (1):
- TUTH, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Yes
supplementary tables will be shared
Supporting Information: Study Protocol
Time Frame: once the study is published
Access Criteria: open

REFERENCES:
- [Background] Gurbuz H, Demir N. Anxiety and Depression Symptoms of Family Members of Intensive Care Unit Patients: A Prospective Observational Study and the Lived Experiences of the Family Members. Avicenna J Med. 2023 Jun 16;13(2):89-96. doi: 10.1055/s-0043-1769933. eCollection 2023 Apr. PMID 37435558
- [Background] Pochard F, Azoulay E, Chevret S, Lemaire F, Hubert P, Canoui P, Grassin M, Zittoun R, le Gall JR, Dhainaut JF, Schlemmer B; French FAMIREA Group. Symptoms of anxiety and depression in family members of intensive care unit patients: ethical hypothesis regarding decision-making capacity. Crit Care Med. 2001 Oct;29(10):1893-7. doi: 10.1097/00003246-200110000-00007. PMID 11588447
- [Background] Kulkarni HS, Kulkarni KR, Mallampalli A, Parkar SR, Karnad DR, Guntupalli KK. Comparison of anxiety, depression, and post-traumatic stress symptoms in relatives of ICU patients in an American and an Indian public hospital. Indian J Crit Care Med. 2011 Jul;15(3):147-56. doi: 10.4103/0972-5229.84891. PMID 22013306
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Risal A, Manandhar K, Linde M, Koju R, Steiner TJ, Holen A. Reliability and Validity of a Nepali-language Version of the Hospital Anxiety and Depression Scale (HADS). Kathmandu Univ Med J (KUMJ). 2015 Apr-Jun;13(50):115-24. doi: 10.3126/kumj.v13i2.16783. PMID 26657079
- [Background] Bialek K, Sadowski M. Stress, anxiety, depression and basic hope in family members of patients hospitalised in intensive care units - preliminary report. Anaesthesiol Intensive Ther. 2021;53(2):134-140. doi: 10.5114/ait.2021.105728. PMID 34006051